CLINICAL TRIAL: NCT01152918
Title: TLC-Plus: A Study to Evaluate the Feasibility of an Enhanced Test, Link to Care, Plus Treat Approach for HIV Prevention in the United States
Brief Title: Evaluating Methods to Increase HIV Testing, Access to HIV Care, and HIV Prevention Strategies
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: HIV Prevention Trials Network (Network)
Collaborators: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HPTN 065; 1U01AI068619 (NIH)
Record Dates: First submitted 2010-06-28; First posted 2010-06-29 (Estimated); Last update posted 2025-04-01 (Actual); Status verified 2025-03

CONDITIONS: HIV Infection
Keywords: HIV Prevention; HIV Treatment; HIV Test and Treat Model of Prevention; ART for Prevention; Prevention for HIV Positives; Financial Incentives; Computer-delivered risk-reduction counseling
MeSH Terms: conditions — HIV Infections

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (6):
- Linkage-to-Care Component: Financial Incentive (FI) (Experimental): Provide financial incentives for linkage to HIV care.
  Interventions: Behavioral: Linkage-to-Care Component: Financial Incentive (FI)
- Linkage-to-Care Component: Standard of Care (SOC) (Active Comparator): Provide the SoC to patients for linkage to HIV care
  Interventions: Behavioral: Linkage-to-Care Component: Standard of Care (SOC)
- Viral Suppression Component: FI (Experimental): Provide financial incentives for viral load suppression
  Interventions: Behavioral: Viral Suppression Component: FI
- Viral Suppression Component: SOC (Active Comparator): Provide the SoC to patients for viral load suppression
  Interventions: Behavioral: Viral Suppression Component: SOC
- Prevention for Positives Component: Intervention (Experimental): Computerized HIV risk reduction counseling program
  Interventions: Behavioral: Prevention for Positives Component: Counseling and SOC
- Prevention for Positives Component: SOC (Active Comparator): Receive SOC for HIV infection
  Interventions: Behavioral: Prevention for Positives Component: SOC

INTERVENTIONS:
Behavioral: Linkage-to-Care Component: Financial Incentive (FI) — Test sites assigned to this arm will provide coupons to all people who are found to be HIV-infected after testing and who are not already linked to HIV care. The coupons can be redeemed at a participating HIV care site for gift cards.
  Arms: Linkage-to-Care Component: Financial Incentive (FI)
Behavioral: Linkage-to-Care Component: Standard of Care (SOC) — Each person who receives an HIV positive test result, and is not currently in care, will be directed to HIV care sites using the site's SOC procedures.
  Arms: Linkage-to-Care Component: Standard of Care (SOC)
Behavioral: Viral Suppression Component: FI — HIV-infected participants who are receiving ART will be offered FIs upon the confirmation of each suppressed viral load measurement (less than 400 copies/mL).
  Arms: Viral Suppression Component: FI
Behavioral: Viral Suppression Component: SOC — HIV-infected participants who are receiving ART will be offered support via the site's SOC procedures to attend HIV care site visits and remain adherent to their ART regimen in order to achieve and maintain viral load suppression.
  Arms: Viral Suppression Component: SOC
Behavioral: Prevention for Positives Component: Counseling and SOC — Participants will complete a computer-delivered counseling program that emphasizes HIV prevention strategies for HIV-infected people.
  Arms: Prevention for Positives Component: Intervention
Behavioral: Prevention for Positives Component: SOC — Participants will receive SOC from their HIV care site.
  Arms: Prevention for Positives Component: SOC

SUMMARY:
This is a five-part study that will take place in the Bronx, New York (NY), and Washington, District of Columbia (DC). The different components of the study will focus on increasing the number of people being tested for HIV, evaluating ways to link HIV-infected people to HIV care sites, evaluating methods to reinforce antiretroviral therapy (ART) adherence, and evaluating a counseling program that focuses on HIV prevention. (Details for only three components of this study are included in ClinicalTrials.gov (Linkage-to-Care, Viral Suppression and Prevention for Positives) because they are the only ones that were randomized and had prescriptive interventions.)

DETAILED DESCRIPTION:
The five components of the study include the following:

Expanded HIV Testing: The purpose of this part of the study is to increase the number of people being tested for HIV. In select study sites in the Bronx, NY, and Washington, D.C., HIV testing will be expanded in emergency departments (EDs) and upon hospital admission. The study will provide additional resources to expand outreach and marketing efforts in these communities. This part of the study will take place over 36 months.

Linkage-to-Care: This part of the study will take place over a 24-month period. The purpose is to compare the effectiveness of a financial incentive (FI) program to link HIV-infected people from HIV test sites to HIV care sites versus standard of care (SOC). Each HIV test site will be randomly assigned to either the FI program or SOC. At the FI sites, people who receive an HIV positive test result will receive a coupon that can be redeemed for gift cards at participating HIV care sites.

Viral Suppression: This part of the study will assess the effectiveness of an FI program at helping HIV-infected people achieve and maintain a viral load of less than 400 copies/mL compared to SOC. Each HIV care site will be randomly assigned to either the FI program or SOC. At the FI sites, HIV-infected people will receive gift cards if their viral load remains below 400 copies/mL. People are eligible to receive FIs once every 3 months throughout the 24-month study period.

Prevention for Positives: The purpose of this component of the study is to evaluate the effectiveness of a computer-delivered counseling program that focuses on HIV risk reduction behaviors for HIV-infected people. Participants will be randomly assigned to the counseling program and SOC or SOC alone. All participants will answer questions on the computer about HIV testing and care at baseline and Months 3, 6, 9, 12, and 18. Study researchers will review participants' medical records at study entry and every 3 months up to Month 18.

Survey of Patients and Providers: Participants in the Prevention for Positives component of the study will complete a computerized survey at the baseline and Month 12 visit, which will assess knowledge and attitudes about ART. Health care providers at the HIV care sites will complete Web-based surveys before and after the Viral Suppression component of the study.

ELIGIBILITY:
Inclusion/Exclusion Criteria for Linkage-to-Care Component:

The Linkage-to-Care component of the study will include all individuals ages 12 and older who are permitted to consent, or can be consented for HIV care by a parent/legal guardian according to New York State or Washington, D.C. law, and who are newly found to be HIV-positive at HIV test sites participating in the study. This study component will also include individuals who have been previously diagnosed with HIV but have been out of care for at least a year and are reconfirmed for HIV infection by standard laboratory tests

Inclusion/Exclusion Criteria for Viral Suppression Component:

The study population for the viral suppression component of the study will include all individuals ages 12 and older who are permitted to consent, or can be consented for HIV care by a parent/legal guardian according to New York State or Washington, D.C. law, who have initiated care at participating HIV care sites.

Inclusion Criteria for Prevention for Positives Component:

* All people who are permitted to consent for HIV care according to New York State or Washington, D.C. law
* Receiving care at the selected HIV care sites in the Bronx or Washington, D.C.
* Have attended the clinic one or more times in the 7 months before study entry
* Able to understand either spoken English or Spanish
* Able and willing to provide informed consent
* Participants enrolled into the Prevention for Positives component of the study will participate in the Patient Survey Component

Exclusion Criteria for Prevention for Positives Component:

* Not seen in the clinic in the 7 months before study entry
* History or evidence of altered mentation, inebriation, or substance use that would interfere with participation in the study
* Unable or unwilling to provide informed consent
* Participation in another study focusing on HIV prevention for positives

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 18442 (Actual)
Dates: Start 2010-09; Primary Completion 2014-12 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
Expanded HIV Testing Component: Number and results of HIV tests per month in publicly funded testing sites (local health department data) | Measured at Month 36
Expanded HIV Testing Component: Number, transmission category, and testing source of newly identified cases in HIV surveillance data | Measured at Month 36
Expanded HIV Testing Component: Initial CD4 cell count of newly identified HIV cases in surveillance data | Measured at Month 36
Expanded HIV Testing Component: Number of newly identified HIV cases concomitantly diagnosed with AIDS in surveillance data | Measured at Month 36
Expanded HIV Testing Component: Proportion of persons in the community tested for HIV in the last year (local population-based behavioral surveys) | Measured at Month 36
Expanded HIV Testing Component: Proportion and number of total ED visits and admissions to hospital where patients receive HIV testing | Measured at Month 36
Expanded HIV Testing Component: Number of HIV tests in EDs where HIV infection is newly identified | Measured at Month 36
Expanded HIV Testing Component: Number of HIV tests in hospital admissions where patients receive HIV testing | Measured at Month 36
Expanded HIV Testing Component: Proportion of hospital admissions who have newly identified HIV infection | Measured at Month 36
Expanded HIV Testing Component: Number of tested patients identified with previously diagnosed HIV who are not in care | Measured at Month 36
Expanded HIV Testing Component: Cost of support for additional staff and HIV tests | Measured at Month 36
Linkage-to-Care Component: Number of individuals eligible for incentives and number of individuals receiving incentives (upon linkage to HIV care) at participating sites | Measured at Month 24
Linkage-to-Care Component: Cost of the program, including staffing, infrastructure, and incentives | Measured at Month 24
Linkage-to-Care Component: Proportion of HIV-infected people at each site with newly detected HIV infection or who were previously diagnosed but were out of care, and who are presently linked to care | Measured at Month 24
Linkage-to-Care Component: Mean time interval at each site from HIV diagnosis (Western Blot confirmation) to first CD4 cell count or viral load for those with newly detected HIV infection and those who were previously diagnosed but were out of care | Measured at Month 24
Linkage-to-Care Component: Proportion of HIV-infected people at a testing site with at least two CD4 cell count and viral load measurements in the prior year | Measured at Month 24
Viral Suppression Component: Number of individuals eligible for incentives and receiving incentives at a select subset of sites for select time points | Measured at Month 24
Viral Suppression Component: Cost of program, including staffing, infrastructure, and incentives | Measured at Month 24
Viral Suppression Component: Probability of an HIV-infected patient in care at a site having a suppressed viral load (less than 400 copies/mL) in the 12-month calendar assessment period beginning 12 months after initiation of the assessment period | Measured at Month 24
Viral Suppression Component: Number of identified HIV-infected patients in care who have sustained viral suppression | Measured at Month 24
Prevention for Positives Component: Proportion of participants reporting any unprotected vaginal or anal sex in the previous 3 months | Measured at Month 12 and 18

SECONDARY OUTCOMES:
Prevention for Positives Component: Number of sex partners of discordant or unknown HIV status with whom participant had unprotected vaginal or anal sex in the previous 3 months | Measured at Month 12 and 18
Prevention for Positives Component: Number of sex partners with whom the participant had unprotected sex in the previous 3 months | Measured at Month 12 and 18
Prevention for Positives Component: Number of persons with whom the participant shared needles after self use in the previous 3 months | Measured at Month 12 and 18

CONTACTS AND LOCATIONS:
Overall Officials: Wafaa El-Sadr, MD, MPH, Study Chair — Columbia University and Harlem Hospital; Bernard Branson, MD, Study Chair — Centers for Disease Control and Prevention
Locations (2):
- United States (2):
  - DC clinics, Washington D.C., District of Columbia
  - Bronx clinics, New York, New York

REFERENCES:
- [Background] El-Sadr WM, Affrunti M, Gamble T, Zerbe A. Antiretroviral therapy: a promising HIV prevention strategy? J Acquir Immune Defic Syndr. 2010 Dec;55 Suppl 2(Suppl 2):S116-21. doi: 10.1097/QAI.0b013e3181fbca6e. PMID 21406980
- [Background] London AJ, Borasky DA Jr, Bhan A; Ethics Working Group of the HIV Prevention Trials Network. Improving ethical review of research involving incentives for health promotion. PLoS Med. 2012;9(3):e1001193. doi: 10.1371/journal.pmed.1001193. Epub 2012 Mar 27. PMID 22479154
- [Background] El Sadr W, Branson BM, Donnell DJ; Hall HI, Gamble TR, Farrior JH, Watkins PS, Greene E, Zerbe A, Buchacz K, Kurth A. TLC-Plus (HPTN 065): Test, Link to Care Plus Treat HPTN 065. (Oral Presentation). 2nd International HIV Treatment as Prevention Workshop, Vancouver BC; April 24, 2012
- [Background] King GM, Sista N, Richards-Clarke C, Turner M, Gamble T, Lucas J. Community Engagement for HPTN 065 (TLC-Plus) study, a community-based study evaluating the feasibility of a combination of interventions to prevent HIV transmission in the US. Poster at the XIX International AIDS Conference, Washington, DC: July 24, 2012. TUPE411.
- [Background] Donnell DJ, Hall HI, Gamble T, Beauchamp G, Griffin AB, Torian LV, Branson B, El-Sadr WM. Use of HIV case surveillance system to design and evaluate site-randomized interventions in an HIV prevention study: HPTN 065. Open AIDS J. 2012;6:122-30. doi: 10.2174/1874613601206010122. Epub 2012 Sep 7. PMID 23049660
- [Background] Adamson B, Donnell D, Dimitrov D, Garrison L, Beauchamp G, Gamble T, Branson B, El Sadr W. The Cost Effectiveness of the Financial Incentives intervention for Viral Suppression in HPTN 065. Poster 1045 at CROI 2017, Seattle, WA: February 16, 2017, Session P-X4
- [Result] Greene E, Buchacz K, Gamble T, Beauchamp G, McKinstry L, Wood A, Telzak E, Branson B, El-Sadr W. Linkage-to-Care and ART Adherence Practices at Participating Sites in HPTN 065 (TLC-Plus) Study. Poster at the XIX International AIDS Conference, Washington, DC: July 26, 2012. THPE120
- [Result] Gray KM, Branson B, Donnell DJ, Beauchamp G, Hu X, Wang Z, El Sadr W, Hall HI. HIV testing in six cities using behavioral surveillance data for the TLC-Plus (HPTN 065) study. Poster at the XIX International AIDS Conference, Washington, DC: July 24, 2012. TUPE293.
- [Result] Donnell DJ, Hall HI, Beauchamp G, Gray KM, Griffin AB, Brady KA, Meyer J, Benbow N, Torian LV, Branson B, El Sadr W. Assessing viral suppression amongst HIV patients accessing care in five cities using US HIV surveillance data for the TLC-Plus (HPTN 065) study. Poster at the XIX International AIDS Conference, Washington, DC: July 25, 2012. WEPE115.
- [Result] Greene E, Taylor J, Pack A, Stanton J, Shelus V, Tolley E, D'Angelo L, El-Sadr W, and Gamble T. Understanding of Viral Load among Participants Receiving Financial Incentives for ART Adherence: Findings from a Qualitative Substudy of HPTN 065. Poster at HIV R4P 2014, Cape Town, South Africa: October 29, 2014. A-671-0004-00749. Poster P06.04.
- [Result] Pack A, Stanton J, Greene E, Taylor J, Shelus V, Tolley EE, Brown ST, El-Sadr W, and Gamble T. Unanticipated Impact of Financial Incentives on HIV Patients and Providers: Findings from a Qualitative Substudy (HPTN 065). Poster at HIV R4P 2014, Cape Town, South Africa: October 29, 2014. A-671-0004-00774. Poster P06.02.
- [Result] Pack A, Stanton J, Greene E, Taylor J, Shelus V, Tolley E, Rakhmanina N, El-Sadr W, and Gamble T. Acceptability of Financial Incentives for HIV Viral Suppression: A Qualitative Substudy of HPTN 065. Poster at HIV R4P 2014, Cape Town, South Africa: October 29, 2014. A-671-0005-00765, Poster P23.14.
- [Result] Greene E, Gamble T, Tolley E, Pack A, Stanton J, Taylor J, Shelus V, Leider J, El- Sadr W, and Branson B. The Impact of Implementing a Financial Incentive Program for Viral Suppression on the Clinic Environment: Findings from a Qualitative Substudy of HPTN 065. Poster at HIV R4P 2014, Cape Town, South Africa: October 29, 2014. A-671-0026-00085, Poster P06.03.
- [Result] Gamble T, Corcoran P, Stanton J, Watkins P, Greene E, Farrior J, Elion R, Amenichi-Enahoro S, and El-Sadr W. Geographic Utilization of Gift Cards Used for Financial Incentives to Encourage Viral Suppression: Findings from HPTN 065. Poster at HIV R4P 2014, Cape Town, South Africa: October 29, 2014. A-671-0030-00852, Poster P52.04.
- [Result] Kurth AE, Mayer K, Beauchamp G, McKinstry L, Farrior J, Buchacz K, Donnell D, Branson B, El-Sadr W; HPTN (065) TLC-Plus Study Team. Clinician practices and attitudes regarding early antiretroviral therapy in the United States. J Acquir Immune Defic Syndr. 2012 Dec 15;61(5):e65-9. doi: 10.1097/QAI.0b013e31826a184c.. PMID 23183150
- [Result] El-Sadr W, Branson B, Hall HI, Beauchamp G, Donnell D, Torian L, Zingman B, Lum G, Elion R, Gamble T. Effect of Financial Incentives on Linkage to Care and Viral Suppression: HPTN 065. Oral presentation at CROI 2015, Seattle, Washington: February 24, 2015. Oral abstract 29, Session O-1.
- [Result] Buchacz K, Branson B, Farrior J, Beauchamp G, McKinstry L, Donnell D, Kurth A, Zingman B, Gordin F, El-Sadr W. Providers' Attitudes and Practices Related to ART Use for HIV Care and Prevention. Poster at CROI 2015, Seattle, Washington: February 25, 2015. Poster 1095, Session P-Y2.
- [Result] Chavez P, Buchacz K, Ethridge S, Branson B, Greene E, Gamble T, McKinstry L, Beauchamp G, Connor M, El-Sadr W. Expanding HIV Testing in Hospital Emergency Departments and Inpatient Admissions. Poster 1100 at CROI 2015, Seattle, Washington: February 25, 2015, Session P-Y3.
- [Result] Greene E, Hanscom B, Gamble T, Buchacz K, Jennings A, Naab T, Belloise R, El-Sadr W, Branson B. Evaluation of Process Indicators for Expanded HIV Testing at Hospitals in HPTN 065. Poster CP63 at NHPC 2015, Atlanta, GA: December 8, 2015, Session B.
- [Result] Schackman BR, Eggman AA, Leff JA, Braunlin M, Felsen UR, Fitzpatrick L, Telzak EE, El-Sadr W, Branson BM. Costs of Expanded Rapid HIV Testing in Four Emergency Departments. Public Health Rep. 2016 Jan-Feb;131 Suppl 1(Suppl 1):71-81. doi: 10.1177/00333549161310S109. PMID 26862232
- [Result] El-Sadr WM, Kurth A, Farrior J, Buchacz K, Hansom B, McKinstry L, Elion R, Patel V, Donnell D, Branson B. Prevention for HIV-infected Persons in HPTN 065: Room for Improvement. Poster 989 at CROI 2016, Boston, MA: February 24, 2016, Session P-X4.
- [Result] McKinstry LA, Zerbe A, Hanscom B, Farrior J, Kurth AE, Stanton J, Li M, Elion R, Leider J, Branson B, El-Sadr WM. A Randomized-Controlled Trial of Computer-based Prevention Counseling for HIV-Positive Persons (HPTN 065). J AIDS Clin Res. 2017 Jul;8(7):714. doi: 10.4172/2155-6113.1000714. Epub 2017 Jul 26. PMID 28966842
- [Result] Farrior J, Zerbe A, Kurth A, Hanscom B, McKinstry L, Zingman BS, Gordin F, Donnell D, Branson B, El-Sadr WM. Clinician and Patient Attitudes toward Financial Incentives for HIV care (HPTN 065). Poster 1038 at CROI 2016, Boston, MA: February 25, 2016, Session P-X8.
- [Result] Beauchamp G, El Sadr W, and Donnell D. A Cluster Randomized Analysis of Site-Level HIV Surveillance Data in HPTN 065 (TLC-Plus) Study. Society of Clinical Trials 2016 (May 15-17, 2016)
- [Result] Buchacz K, Farrior J, Beauchamp G, McKinstry L, Kurth AE, Zingman BS, Gordin FM, Donnell D, Mayer KH, El-Sadr WM, Branson B; HPTN 065 Study Team. Changing Clinician Practices and Attitudes Regarding the Use of Antiretroviral Therapy for HIV Treatment and Prevention. J Int Assoc Provid AIDS Care. 2017 Jan/Feb;16(1):81-90. doi: 10.1177/2325957416671410. Epub 2016 Oct 5. PMID 27708115
- [Result] Tolley E, Taylor J, Pack A, Greene E, Stanton J, El-Sadr W, and Gamble T. Role of Financial Incentives along the ART Adherence Continuum: A Qualitative Analysis from the HPTN 065 (TLC-Plus) Study. HIV Research for Prevention 2016 (October 17-21, 2016). Chicago, IL. P15.05.
- [Result] Donnell D, Grey KM, Li J, Wu B, Benbow N, Schuette S, Brady K, Torian L, Xia Q, Callaway BS, Opoku J, Lum G, Meyer J, Hanscom B, Hall I. Encouraging Trends in HIV Diagnoses, Care and Viral Suppression in 5 US Cities, 2009 - 2013: Surveillance-based data from HPTN065 (TLC-Plus). HIV Research for Prevention 2016 (October 17-21, 2016). Chicago, IL. P09.06.
- [Result] Greene E, Pack A, Stanton J, Shelus V, Tolley EE, Taylor J, El Sadr WM, Branson BM, Leider J, Rakhmanina N, Gamble T. "It Makes You Feel Like Someone Cares" acceptability of a financial incentive intervention for HIV viral suppression in the HPTN 065 (TLC-Plus) study. PLoS One. 2017 Feb 9;12(2):e0170686. doi: 10.1371/journal.pone.0170686. eCollection 2017. PMID 28182706
- [Derived] Donnell D. Practical issues in operationalizing the design and outcome evaluation of cluster randomized trials. Clin Trials. 2022 Aug;19(4):407-415. doi: 10.1177/17407745221087465. Epub 2022 Apr 8. PMID 35393864
- [Derived] El-Sadr WM, Donnell D, Beauchamp G, Hall HI, Torian LV, Zingman B, Lum G, Kharfen M, Elion R, Leider J, Gordin FM, Elharrar V, Burns D, Zerbe A, Gamble T, Branson B; HPTN 065 Study Team. Financial Incentives for Linkage to Care and Viral Suppression Among HIV-Positive Patients: A Randomized Clinical Trial (HPTN 065). JAMA Intern Med. 2017 Aug 1;177(8):1083-1092. doi: 10.1001/jamainternmed.2017.2158. PMID 28628702
- See also: TLC-Plus (HPTN 065): Test, Link to Care Plus Treat HPTN 065. (Oral Presentation). 2nd International HIV Treatment as Prevention Workshop, Vancouver BC; April 24, 2012 — https://www.youtube.com/watch?v=yYrlMLb9FTs
- See also: Linkage-to-Care and ART Adherence Practices at Participating Sites in HPTN 065 (TLC-Plus) Study. Poster at the XIX International AIDS Conference, Washington, DC: July 26, 2012. THPE120 — https://www.hptn.org/sites/default/files/inline-files/THPE120_065EGreene.pdf
- See also: Community Engagement for HPTN 065 study, a community-based study evaluating the feasibility of a combination of interventions to prevent HIV transmission in the US. Poster at the XIX International AIDS Conference, Washington, DC: July 24, 2012. — https://www.hptn.org/sites/default/files/inline-files/TUPE411_065GKing.pdf
- See also: HIV testing in six cities using behavioral surveillance data for the TLC-Plus (HPTN 065) study. Poster at the XIX International AIDS Conference, Washington, DC: July 24, 2012. TUPE293. — https://www.hptn.org/sites/default/files/inline-files/TUPE293_065KGray.pdf
- See also: Assessing viral suppression amongst HIV patients accessing care in six cities using US HIV surveillance data for the TLC-Plus (HPTN 065) study. Poster at the XIX International AIDS Conference, Washington, DC: July 25, 2012. WEPE115. — https://www.hptn.org/sites/default/files/inline-files/WEPW115_065DDonnell.pdf
- See also: Understanding of Viral Load among Participants Receiving Financial Incentives for ART Adherence: Findings from a Qualitative Substudy of HPTN 065. Poster at HIV R4P 2014, Cape Town, South Africa: October 29, 2014. A-671-0004-00749. Poster P06.04. — https://www.hptn.org/sites/default/files/2016-05/R4Punderstandingviral.pdf
- See also: Unanticipated Impact of Financial Incentives on HIV Patients and Providers: Findings from a Qualitative Substudy (HPTN 065). Poster at HIV R4P 2014, Cape Town, South Africa: October 29, 2014. A-671-0004-00774. Poster P06.02. — https://www.hptn.org/sites/default/files/2016-05/R4Punanticipated.pdf
- See also: Acceptability of Financial Incentives for HIV Viral Suppression: A Qualitative Substudy of HPTN 065. Poster at HIV R4P 2014, Cape Town, South Africa: October 29, 2014. A-671-0005-00765, Poster P23.14. — https://www.hptn.org/sites/default/files/2016-05/R4Pacceptabilityvs.pdf
- See also: The Impact of Implementing a Financial Incentive Program for VS on the Clinic Environment: Findings from a Qualitative Substudy of HPTN 065. Poster at HIV R4P 2014, Cape Town, South Africa: October 29, 2014. A-671-0026-00085, Poster P06.03. — https://www.hptn.org/sites/default/files/2016-05/R4Pimpactincentives.pdf
- See also: Geographic Utilization of Gift Cards Used for Financial Incentives to Encourage Viral Suppression: Findings from HPTN 065. Poster at HIV R4P 2014, Cape Town, South Africa: October 29, 2014. A-671-0030-00852, Poster P52.04. — https://www.hptn.org/sites/default/files/2016-05/R4Pgiftcarduse.pdf
- See also: Effect of Financial Incentives on Linkage to Care and Viral Suppression: HPTN 065. Oral presentation at CROI 2015, Seattle, Washington: February 24, 2015. Oral abstract 29, Session O-1 — http://www.croiwebcasts.org/console/player/25546?mediaType=audio&
- See also: Providers' Attitudes and Practices Related to ART Use for HIV Care and Prevention. Poster at CROI 2015, Seattle, Washington: February 25, 2015. Poster 1095, Session P-Y2. — https://www.hptn.org/sites/default/files/2016-05/CROI15Providers.pdf
- See also: Expanding HIV Testing in Hospital Emergency Departments and Inpatient Admissions. Poster 1100 at CROI 2015, Seattle, Washington: February 25, 2015, Session P-Y3. — https://www.hptn.org/sites/default/files/2016-05/CROI15EHT.pdf
- See also: Prevention for HIV-infected Persons in HPTN 065: Room for Improvement. Poster 989 at CROI 2016, Boston, MA: February 24, 2016, Session P-X4. — https://www.hptn.org/sites/default/files/2016-05/Poster989_Abstract%2016-643_0.pdf
- See also: Computer-based Prevention Counseling for HIV-infected Persons (HPTN 065). Poster 997 at CROI 2016, Boston, MA: February 24, 2016, Session P-X4. — https://www.hptn.org/sites/default/files/2016-05/Poster997_Abstract%2016-731_0.pdf
- See also: Clinician and Patient Attitudes toward Financial Incentives for HIV care (HPTN 065). Poster 1038 at CROI 2016, Boston, MA: February 25, 2016, Session P-X8. — https://www.hptn.org/sites/default/files/2016-05/Poster1038_Abstract%2016-377_0.pdf